CLINICAL TRIAL: NCT04738448
Title: Examining the Effects of Art Therapy in Reducing Burnout in Healthcare Using the Maslach Burnout Inventory
Brief Title: Examining the Effects of Art Therapy in Reducing Burnout in Healthcare Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Marie Doll, Senior Art Therapist, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00095937
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Burnout, Professional
Keywords: Art Therapy
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art Therapy Group (Experimental)
  Interventions: Behavioral: Art Therapy Group

INTERVENTIONS:
Behavioral: Art Therapy Group — The art therapy intervention will be executed by the same Medical University of South Carolina (MUSC) board-certified art therapist for each group. The art therapist is a masters-level, licensed practitioner who has experience working in the healthcare system and treating providers. The same art therapy practices that are utilized in daily practice at MUSC will be employed in this study, with a focus on reducing burnout symptoms. Pilot testing of the intervention has been performed informally at MUSC with positive feedback reported by healthcare providers.

SUMMARY:
In this study, the investigators aim to examine the effects of art therapy in reducing burnout in healthcare providers. Using the Maslach Burnout Inventory Human Services Survey for Medical Personnel, the investigators will measure burnout in Medical University of South Carolina (MUSC) providers before and after the administration of a 4-week art therapy group.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Employed at MUSC as a healthcare provider
* Able and willing to participate in all 4 art therapy sessions

Exclusion Criteria:

* Individual does not provide direct patient care at MUSC
* Individual works in the same department as the art therapist
* Inability or unwillingness of subject to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Burnout Symptoms | At start of therapy sessions and 4 weeks after therapy sessions
  Measuring burnout symptoms utilizing the Maslach Burnout Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Marie Doll, MA, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No